CLINICAL TRIAL: NCT02536105
Title: Pharmacokinetic Pharmacodynamic Studies of Methylphenidate Extended Release Products in Pediatric Attention Deficit Hyperactivity Disorder
Brief Title: PK/PD Pediatric ADHD Classroom Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); Center for Psychiatry And Behavioral Medicine Inc. (Industry)
Responsible Party: Principal Investigator, Thomas J. Spencer, MD, Associate Chief, Clinical and Research Program, Pediatric Psychopharmacology, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015P001113; 5U01FD005240 (FDA)
Record Dates: First submitted 2015-08-24; First posted 2015-08-31 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Suspensions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Methylphenidate HCl ER tablets 1 (Active Comparator): During the open-label optimization phase, one of the methylphenidate hydrochloride extended-release products will be titrated at weekly intervals of 18mg increments until an optimal dose is achieved or a maximum of 72mg per day is reached. During the double-blind phase, participants will receive blinded treatment each week. The dose of each methylphenidate hydrochloride extended-release product will be determined by the optimized dose during the open-label optimization phase
  Interventions: Drug: Methylphenidate HCl ER tablets 1
- Placebo (Placebo Comparator): During the double-blind period, in one of the 4 study weeks, the study participant will take a blinded placebo instead of one of the the 3 active comparators.
  Interventions: Drug: Placebo
- Methylphenidate HCl ER tablets 2 (Active Comparator): During the open-label optimization phase, one of the methylphenidate hydrochloride extended-release products will be titrated at weekly intervals of 18mg increments until an optimal dose is achieved or a maximum of 72mg per day is reached. During the double-blind phase, participants will receive blinded treatment each week. The dose of each methylphenidate hydrochloride extended-release product will be determined by the optimized dose during the open-label optimization phase
  Interventions: Drug: Methylphenidate HCl ER tablets 2
- Methylphenidate HCl ER for suspension (Active Comparator): During the open-label optimization phase, one of the methylphenidate hydrochloride extended-release products will be titrated at weekly intervals of 18mg increments until an optimal dose is achieved or a maximum of 72mg per day is reached. During the double-blind phase, participants will receive blinded treatment each week. The dose of each methylphenidate hydrochloride extended-release product will be determined by the optimized dose during the open-label optimization phase
  Interventions: Drug: Methylphenidate HCl ER for suspension

INTERVENTIONS:
Drug: Methylphenidate HCl ER tablets 1
  Arms: Methylphenidate HCl ER tablets 1
Drug: Placebo
  Arms: Placebo
Drug: Methylphenidate HCl ER tablets 2
  Arms: Methylphenidate HCl ER tablets 2
Drug: Methylphenidate HCl ER for suspension
  Arms: Methylphenidate HCl ER for suspension

SUMMARY:
The purpose of this study is to evaluate the association between blood drug levels and the corresponding scores of commonly used behavioral instruments based upon data collected following administration of three different methylphenidate hydrochloride extended-release drug products in children with ADHD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, 4-treatment and 4-period crossover study conducted in a school laboratory environment to evaluate the hour-by-hour behavioral instrument scores and hour-by-hour PK of 3 different extended-release MPH formulations as well as placebo in children with ADHD. The complete study consists of three periods: Screening, Dose Titration and Double-Blind Crossover in a Laboratory Classroom.

The double-blind phase will consist of four periods (or four weeks): each week will consist of blinded administration with one of the three active methylphenidate hydrochloride treatments or placebo from Sunday through Saturday. On the last day of each period (Saturday), study participants will be evaluated in a laboratory classroom setting. On Saturdays, the blinded doses of each study drug will be administered at the school site by study staff on the morning of the test laboratory classroom day. On the other days, the medication will be taken in the morning at home.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients
2. Ages 6-12 years at time of screening
3. Judged by the investigator to be physically healthy and suitable for participation in the study
4. Diagnosis of DSM-5ADHD combined, predominantly inattentive or hyperactive/impulsive presentation, per clinical evaluation and confirmed by the MINI-KID
5. Clinical Global Impressions-Severity (CGI-S) ≥ 3
6. ≥ 90th percentile normative value for gender and age on the ADHD RS-IV total score at screening or baseline
7. Study participant has a parent/legal guardian who is willing and able to give written informed consent for him/her to participate in the study
8. Study participant must be able to give assent to participate in the trial
9. Study participant and legal guardian must be able to speak and understand English
10. Able to tolerate multiple finger pricks
11. Willing to comply with all study procedures

Exclusion Criteria:

1. Current (last month) psychiatric diagnosis other than specific phobia, motor skills disorders, oppositional defiant disorder, sleep disorders, elimination disorders, adjustment disorders, learning disorders, or communication disorders. Participants with school phobia or separation anxiety will not be eligible
2. Cognitively impaired, in the investigator's opinion
3. Any clinically significant chronic medical condition that, in the judgment of the investigator, may interfere with the participant's ability to participate in the study
4. Seizure disorder excluding a history of febrile seizures
5. Thyroid disease
6. Tourette's disorder or chronic tic disorder (mild medication induced tics are allowed)
7. Serious cardiac condition including cardiomyopathy, serious arrhythmias, structural cardiac disorders, or severe hypertension
8. Glaucoma
9. Current or recent (within the past 6 months) DSM-5 drug dependence or substance abuse (excluding nicotine and caffeine)
10. Pregnant or nursing females. Females must have a negative urine pregnancy test at screening as well as four additional visits and must be abstinent or use adequate and reliable contraception throughout the study
11. Currently treated and satisfied with ADHD medication
12. Current psychotropic medications other than sedative hypnotics for sleep
13. Use of atomoxetine, clonidine, guanfacine or a monoamine oxidase inhibitor within 28 days of the baseline visit
14. Participation in another investigational medication study within 30 days prior to screening
15. Clinically significant abnormal laboratory result, electrocardiogram (ECG) result, physical examination, or vital signs at screening that the investigator considers to be inappropriate to allow participation in the study
16. Planned use of prohibited drugs from the baseline visit through the end of the trial
17. History of allergic reaction or a known or suspected sensitivity to any substance that is contained in the study drugs
18. Food allergies that are determined by the PI as too severe to be easily accommodated for during the study
19. Inability to swallow study medication

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 88 individuals signed consent. 82 individuals were eligible for the study. 80 individuals were exposed to the open-label phase (Methylphenidate HCL ER Tablets 1). 76 individuals entered the double-blind phase. 72 individuals completed the entire study. Since this is a crossover study, these were the same individuals (88 consented, not 301).
Groups:
- All Participants: Participants received 4 different medications at the following 5 time points.
  1. Open-label phase MPH ER Tab 1
  2. Crossover Placebo
  3. Crossover MPH ER Tab 1
  4. Crossover MPH ER Tab 2
  5. Crossover MPH ER Suspension
Period: Concerta Open Label
Arm/Group | All Participants
Started | 80
Completion of Phase | 76
Completed (Number of participants who completed the entire study.) | 72
Not Completed | 8
Period: Placebo
Arm/Group | All Participants
Started | 74
Completion of Placebo Day | 74
Completed (Number of participants who completed the entire study.) | 72
Not Completed | 2
Period: Methylphenidate HCl ER Tablet 1
Arm/Group | All Participants
Started | 72
Completion of MPH HCl ER Tab 1 Day | 72
Completed (Number of participants who completed the entire study.) | 72
Not Completed | 0
Period: Methylphenidate HCl ER Tablet 2
Arm/Group | All Participants
Started | 73
Completion of MPH HCl ER Tablet 2 Phase | 73
Completed (Number of participants who completed the entire study.) | 72
Not Completed | 1
Period: Methylphenidate HCl ER Suspension
Arm/Group | All Participants
Started | 74
Completion of MPH HCl ER Susp Phase | 74
Completed (Number of participants who completed the entire study.) | 72
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: 80 individuals were exposed in the open-label phase of the study which involved Methylphenidate HCl ER Tablets 1 (Concerta).
Groups:
- Open-Label: Methylphenidate HCl ER Tablets 1: During the open-label optimization phase, one of the methylphenidate hydrochloride extended-release products will be titrated at weekly intervals of 18mg increments until an optimal dose is achieved or a maximum of 72mg per day is reached.
  Methylphenidate HCl ER tablets 1
Arm/Group | Open-Label: Methylphenidate HCl ER Tablets 1
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 80
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.45 (1.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 45
  More than one race | 16
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Permanent Product Measure of Performance (PERMP) for Three Methylphenidate Hydrochloride Extended-release Drug Products
Description: The Permanent Product Measure of Performance (PERMP) involves objective individualized mathematics tests. Scores will be obtained ten times on each classroom day at pre-dose, and at approximately 0.5, 1.5, 2.5, 4, 5, 6, 8, 10 and 12 hours post-dose. PERMP Attempted is reported here. Scale ranges 0 math questions answered to 400 math questions answered. The more number of questions answered (better score), the higher the PERMP Attempted score is.
Time Frame: 0.5, 1.5, 2.5, 4, 5, 6, 8, 10 and 12 hours post-dose on each classroom day
Population: Note that not all participants who entered the study completed all arms and all time points, hence the discrepancy in number of participants analyzed between arms and different time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Methylphenidate HCl ER Tablets 1: During the open-label optimization phase, one of the methylphenidate hydrochloride extended-release products will be titrated at weekly intervals of 18mg increments until an optimal dose is achieved or a maximum of 72mg per day is reached. During the double-blind phase, participants will receive blinded treatment each week. The dose of each methylphenidate hydrochloride extended-release product will be determined by the optimized dose during the open-label optimization phase
  Methylphenidate HCl ER tablets 1
- Placebo: During the double-blind period, in one of the 4 study weeks, the study participant will take a blinded placebo instead of one of the the 3 active comparators.
  Placebo
- Methylphenidate HCl ER Tablets 2: During the double-blind phase, participants will receive blinded treatment each week. The dose of each methylphenidate hydrochloride extended-release product will be determined by the optimized dose during the open-label optimization phase
  Methylphenidate HCl ER tablets 2
- Methylphenidate HCl ER for Suspension: During the double-blind phase, participants will receive blinded treatment each week. The dose of each methylphenidate hydrochloride extended-release product will be determined by the optimized dose during the open-label optimization phase
  Methylphenidate HCl ER for suspension
Arm/Group | Methylphenidate HCl ER Tablets 1 | Placebo | Methylphenidate HCl ER Tablets 2 | Methylphenidate HCl ER for Suspension
Number analyzed (Participants) | 67 | 72 | 66 | 68
score on a scale
  HOUR 0 | 66.925 (43.7199) | 95.361 (53.7921) | 80.621 (57.0923) | 92.176 (70.6378)
  HOUR .5 | 78.463 (58.8659) | 90.194 (67.6144) | 88.333 (73.9824) | 114.294 (76.9904)
  HOUR 1.5: number analyzed (Participants) | 67 | 71 | 66 | 68
  HOUR 1.5 | 112.493 (62.1631) | 89.366 (74.0415) | 112.364 (70.9701) | 131.191 (65.958)
  HOUR 2.5 | 124.313 (65.4757) | 86.236 (61.5375) | 127.848 (71.7946) | 139.132 (75.4724)
  HOUR 4 | 120.985 (64.1158) | 85.986 (63.3276) | 130.591 (65.7204) | 129.735 (70.0097)
  HOUR 5: number analyzed (Participants) | 67 | 71 | 66 | 67
  HOUR 5 | 103.985 (58.6211) | 71.718 (56.1392) | 117.879 (63.5952) | 122.91 (72.3134)
  HOUR 6: number analyzed (Participants) | 66 | 69 | 65 | 66
  HOUR 6 | 107.303 (64.5355) | 73.42 (48.0843) | 112.985 (68.729) | 124.862 (68.9096)
  HOUR 8: number analyzed (Participants) | 67 | 71 | 66 | 67
  HOUR 8 | 117.403 (66.8252) | 82.408 (59.657) | 123.803 (65.2423) | 97.358 (58.9822)
  HOUR 10: number analyzed (Participants) | 67 | 71 | 66 | 67
  HOUR 10 | 113.03 (65.3686) | 80.761 (60.2045) | 103.864 (60.7101) | 99.881 (66.7032)
  HOUR 12: number analyzed (Participants) | 67 | 71 | 66 | 67
  HOUR 12 | 112.09 (76.5476) | 82.718 (50.4251) | 109.909 (64.7206) | 82.642 (58.0224)

2. Primary Outcome: Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) Rating Scale for Three Methylphenidate Hydrochloride Extended-release Drug Products
Description: The Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) scale is a validated, 13-item rating of subjective impairment of classroom behaviors (0 = normal/no impairment; 1 = slight impairment; 2 = mild impairment; 3 = moderate impairment; 4 = severe impairment; 5 = very severe impairment; 6 = maximal impairment). The SKAMP consists of four subscales: SKAMP-Attention, SKAMP-Deportment, SKAMP-Quality of Work, and SKAMP-Compliance, in addition to SKAMP-Total (reported here). SKAMP-Total is a sum of the four sub-scales and has a range of 0-78. The higher the score, the higher the impairment. Scores will be obtained during each classroom cycle during each full laboratory classroom day at pre-dose, and at 0.5, 1.5, 2.5, 4, 5, 6, 8, 10, and 12 hours post-dose. The scores will be based on the child's behavior during 20 minutes of each cycle.
Time Frame: 0.5, 1.5, 2.5, 4, 5, 6, 8, 10 and 12 hours post-dose on each classroom day
Population: Note that not all participants who entered the study completed all arms. Thus, the number differs between the arms to reflect the number of participants who provided data for that arm. N=67 for all MPH HCl ER tab 1 time points. N=72 for all placebo time points. N=66 for all MPH HCl tab 2 time points. N=68 for all MPH Hcl ER susp timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate HCl ER Tablets 1 | Placebo | Methylphenidate HCl ER Tablets 2 | Methylphenidate HCl ER for Suspension
Number analyzed (Participants) | 67 | 72 | 66 | 68
units on a scale
  HOUR 0 | 36.4328 (13.1209) | 27.7917 (13.475) | 34.2879 (14.4497) | 33.4706 (14.7855)
  HOUR .5 | 35.2836 (15.2204) | 30.7361 (14.8029) | 32.1061 (13.2875) | 27.0588 (16.1466)
  HOUR 1.5 | 23.4328 (15.9917) | 33.9722 (15.354) | 25.4091 (13.8775) | 17.8676 (12.9233)
  HOUR 2.5 | 20.0746 (12.6087) | 33.4861 (13.2399) | 20.3939 (13.4163) | 15.8088 (10.9466)
  HOUR 4 | 19.1642 (12.216) | 33.4028 (13.7888) | 15.7576 (10.5233) | 17.4412 (12.3462)
  HOUR 5 | 22.3881 (12.7588) | 36.2917 (14.1962) | 17.1061 (11.9526) | 20.6765 (13.3108)
  HOUR 6 | 22.1642 (12.8766) | 35.00 (14.7601) | 15.8636 (10.5158) | 22.8382 (14.8078)
  HOUR 8 | 21.0448 (11.8186) | 35.0972 (14.4038) | 19.3788 (12.0509) | 28.3382 (14.6548)
  HOUR 10 | 20.7164 (13.313) | 34.2222 (14.0554) | 24.4394 (15.1679) | 31.9412 (13.7329)
  HOUR 12 | 23.0746 (15.3981) | 32.2778 (14.396) | 27.3485 (15.3508) | 34.7353 (15.3123)

3. Primary Outcome: Maximum Drug Concentration Observed (Cmax) for Three Methylphenidate Hydrochloride Extended-release Drug Products
Description: PK samples will be taken eight times on each classroom day at approximately 0.5, 1.5, 2.5, 4, 5, 6, 8, and 12 hours post-dose, and Cmax will be measured. The objectives of this measure is to estimate PK metrics, including Cmax, appropriate for characterizing rate and extent of absorption in each phase of the drug release and the evaluate the disposition and eliminating processes for each medication studied. The minimum value is pg/mL and there is was no maximum defined prior to the interventions.
Time Frame: 0.5, 1.5, 2.5, 4, 5, 6, 8, and 12 hours post-dose on each classroom day
Population: 76 participants entered the double-blind randomization phase and each participant provided at least one data point for these analyses.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Methylphenidate HCl ER Tablets 1 | Placebo | Methylphenidate HCl ER Tablets 2 | Methylphenidate HCl ER for Suspension
Number analyzed (Participants) | 76 | 76 | 76 | 76
pg/mL | 76339 (55690) | 4327 (4594) | 81611 (46702) | 81498 (66961)

4. Primary Outcome: Time to Reach Cmax (Tmax) for Three Methylphenidate Hydrochloride Extended-release Drug Products
Description: PK samples will be taken eight times on each classroom day at approximately 0.5, 1.5, 2.5, 4, 5, 6, 8, and 12 hours post-dose, and Tmax will be measured
Time Frame: 0.5, 1.5, 2.5, 4, 5, 6, 8, and 12 hours post-dose on each classroom day
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Methylphenidate HCl ER Tablets 1 | Placebo | Methylphenidate HCl ER Tablets 2 | Methylphenidate HCl ER for Suspension
Number analyzed (Participants) | 76 | 76 | 76 | 76
Hours | 7.35 (3.05) | 4.7 (2.99) | 6.35 (2.22) | 3.97 (2.19)

ADVERSE EVENTS:
Time Frame: Baseline (Week 0) to Visit 14 (Week 12) or Drop Visit
Description: Adverse events were collected during the entirety of the study, from consent to completion or withdrawal from the study.
Groups:
- Methylphenidate HCl ER Tablets 2: During the open-label optimization phase, one of the methylphenidate hydrochloride extended-release products will be titrated at weekly intervals of 18mg increments until an optimal dose is achieved or a maximum of 72mg per day is reached. During the double-blind phase, participants will receive blinded treatment each week. The dose of each methylphenidate hydrochloride extended-release product will be determined by the optimized dose during the open-label optimization phase
  Methylphenidate HCl ER tablets 2
- Methylphenidate HCl ER for Suspension: During the open-label optimization phase, one of the methylphenidate hydrochloride extended-release products will be titrated at weekly intervals of 18mg increments until an optimal dose is achieved or a maximum of 72mg per day is reached. During the double-blind phase, participants will receive blinded treatment each week. The dose of each methylphenidate hydrochloride extended-release product will be determined by the optimized dose during the open-label optimization phase
  Methylphenidate HCl ER for suspension
Arm/Group | Methylphenidate HCl ER Tablets 1 | Placebo | Methylphenidate HCl ER Tablets 2 | Methylphenidate HCl ER for Suspension
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/74 | 0/73 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/74 | 0/73 | 0/74
Other Adverse Events (participants affected / at risk) | 69/80 | 12/74 | 20/73 | 23/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate HCl ER Tablets 1 (N=80) | Placebo (N=74) | Methylphenidate HCl ER Tablets 2 (N=73) | Methylphenidate HCl ER for Suspension (N=74)
Insomnia (Psychiatric disorders) | 31 | 1 | 2 | 3
Low Appetite (Gastrointestinal disorders) | 41 | 1 | 4 | 4
Emotional Lability (Psychiatric disorders) | 20 | 2 | 4 | 3 — Emotional Lability, Moodiness, Irritability
Upper Respiratory Infection (Infections and infestations) | 10 | 1 | 1 | 2
GI Distress (Gastrointestinal disorders) | 9 | 3 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 20 | 1 | 3 | 1
Vomited (Gastrointestinal disorders) | 7 | 0 | 2 | 1
Headache (Nervous system disorders) | 16 | 1 | 2 | 3
Anger/Aggression/Oppositional Behavior (Psychiatric disorders) | 6 | 0 | 1 | 0
Dysphoria/Anxiety (Psychiatric disorders) | 2 | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Epistaxis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Ankle Pain/Strain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Strep Throat/Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1
Influenza (Immune system disorders) | 2 | 0 | 0 | 0
Motor Tics (Nervous system disorders) | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0
Bug Bites/Bee Stings (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Otitis Media/Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Carious Teeth (Immune system disorders) | 0 | 0 | 0 | 1
Growth Hormone Deficiency (Endocrine disorders) | 0 | 0 | 0 | 1
Muscle Strain/Pain (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Mouth Ulcers/Bad Breath (Infections and infestations) | 2 | 0 | 0 | 0
Dry Mouth (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Eye Pain (Eye disorders) | 1 | 0 | 0 | 0
Sunburn (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Weight Loss (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Foreign Body Swallowed (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Finger Laceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Flat Affect (Social circumstances) | 2 | 0 | 0 | 0
Urinary Tract Infection (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Toe Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Heart Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Staring Episodes (Psychiatric disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT02536105/Prot_SAP_000.pdf